CLINICAL TRIAL: NCT00686959
Title: Phase 3 Study of Pemetrexed, Cisplatin, and Radiotherapy Followed by Consolidation Pemetrexed Versus Etoposide, Cisplatin, and Radiotherapy Followed by Consolidation Cytotoxic Chemotherapy of Choice in Patients With Unresectable, Locally Advanced, Stage III Non-Small Cell Lung Cancer Other Than Predominantly Squamous Cell Histology
Brief Title: Chemotherapy and Radiation in Treating Participants With Stage 3 Non-Small Cell Lung Cancer
Acronym: PROCLAIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11514; H3E-MC-JMIG (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Etoposide; Vinorelbine; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Pemetrexed + Cisplatin and TRT (Experimental): Participants were treated with Pemetrexed plus Cisplatin and concurrent thoracic radiation therapy (TRT) ("Concurrent Phase") for three 21-day cycles, followed by a 3-5 week "Recovery Period," then treated with consolidation chemotherapy with pemetrexed ("Consolidation Phase") for up to four 21-day cycles
  Concurrent Phase:
  Pemetrexed: 500 milligrams per meter squared (mg/m^2), intravenous (IV) on Day 1 of each 21-day cycle for 3 cycles.
  Cisplatin: 75 mg/m^2, IV on Day 1 of each 21-day cycle x 3 cycles. TRT: Beginning on Day 1 of chemotherapy, once daily fractions (2 Gray [Gy] per day), 5 days a week for 6 weeks and 3 days to target 66 Gy in 33 fractions.
  Consolidation Phase:
  Pemetrexed: 500 mg/m^2, IV on Day 1 of each 21-day cycle up to 4 cycles
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Radiation: Thoracic Radiation Therapy (TRT)
- Arm B: Etoposide + Cisplatin and TRT (Active Comparator): Participants were treated with Etoposide plus Cisplatin and concurrent TRT ("Concurrent Phase") for two 28-day cycles, followed by a 3-5 week "Recovery Period," then received consolidation treatment with cytotoxic chemotherapy of choice ("Consolidation Phase") for up to 2 cycles
  Concurrent Phase:
  Etoposide/Cisplatin (28-day cycle); Etoposide: 50 mg/m^2, IV on Days 1 to 5 and Days 29 to 33 and Cisplatin: 50 mg/m^2, IV on Days1, 8, 29, and 36
  Consolidation Phase options:
  Option 1: Continue the same treatment plan as Concurrent Phase Option 2: Vinorelbine/Cisplatin (21-day cycle); Vinorelbine: 30 mg/m^2, IV on Days 1, 8, 22, and 29; Cisplatin: 75 mg/m^2, IV on Days 1 and 22 Option 3: Paclitaxel/Carboplatin (21-day cycle); Paclitaxel: 200 mg/m^2, IV, on Days 1 and 22; Carboplatin: area under the concentration-time curve (AUC) = 6 (Carboplatin dosing based on calculated creatinine clearance), IV on Days 1 and 22
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Vinorelbine; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Thoracic Radiation Therapy (TRT)

INTERVENTIONS:
Drug: Pemetrexed — infusion over 10 minutes
  Other Names: Alimta; LY231514
  Arms: Arm A: Pemetrexed + Cisplatin and TRT
Drug: Cisplatin — infusion over 60 minutes with adequate anti-emetic treatment and appropriate hydration per local practice guidelines
Drug: Etoposide — administered per local practice guidelines over a minimum of 30 minutes
  Arms: Arm B: Etoposide + Cisplatin and TRT
Drug: Vinorelbine — administered over 6-10 minutes infusion per local practice guidelines
  Arms: Arm B: Etoposide + Cisplatin and TRT
Drug: Paclitaxel — administered as a 3-hour infusion
  Arms: Arm B: Etoposide + Cisplatin and TRT
Drug: Carboplatin — administered per local practice guidelines over 30 minutes
  Arms: Arm B: Etoposide + Cisplatin and TRT
Radiation: Thoracic Radiation Therapy (TRT)

SUMMARY:
This study will compare the overall survival of participants with locally-advanced, Stage III Non-Small Cell Lung Cancer (NSCLC) with nonsquamous cell histology.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have Stage IIIA or IIIIB NSCLC of the non-squamous type
* Participants must have measureable tumor lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines or disease that can be evaluated on computerized tomography (CT) scan
* Participants must be physically mobile, take care of themselves and must be up and about and able to perform light activities, such as light housework or office work
* Participants must be 18 years of age or older
* Participants must have lost no more than 10% of their body weight in the previous 3 months
* Women must be sterile, postmenopausal, or on contraception, and men must be sterile or on contraception
* Participants' test results assessing the function of their blood forming tissue, kidneys, liver, and lungs must be satisfactory
* Participants with Stage IIIB NSCLC who have supraclavicular nodal involvement may be entered into this study. However, participants with cervical nodes are not permitted. The upper border of supraclavicular nodes must not extend above the upper border of the lateral end of the clavicle, extended medially.

Exclusion Criteria:

* Participants cannot have other on-going (uncontrolled) illnesses, including active infections, recent heart problems, or psychiatric illnesses
* Participants who are unable to take vitamins (including injections of vitamin B12) or oral cortisone medication
* Participants who have had a heart attack (myocardial infarction) or other cardiac issues within 6 months of the trial
* Participants who have received other investigational drugs within the last 30 days
* Participants who are unable to stop taking more than 1.3 grams of aspirin on a daily basis or non-steroidal anti-inflammatory agents
* Participants who have diseases considered for surgical treatment as part of their care plan, such as Pancoast or superior sulcus tumors
* Participants who had prior thoracic radiation. However, other prior radiotherapy is allowed. Participants must have recovered from the toxic effects of the treatment prior to study enrollment. Participants may not have received whole pelvis radiation or radiation to more than 25% of their bone marrow. Prior radiotherapy must have been completed at least 30 days prior to study treatment.
* Participants who have a radiation treatment plan that would expose more than 35% of the volume of their lung to 20 gray (Gy) or more of radiation
* Participants who have concurrent cancer from another primary site requiring treatment of any kind within the past 5 years. Exemptions to this will be permitted on a case-by-case basis after prior approval by the Sponsor physician or designate if the investigator believes the participant's risk of recurrence and death is very low. Curatively treated nonmelanoma skin cancer or in situ carcinoma of any origin is allowed. Participants with recurrence of a previously resected lung cancer or who have a second primary lung cancer are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2008-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (133):
- United States (50):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duarte, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fountain Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thomasville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quincy, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Albany, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westwood, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairhaven, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bedford, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longview, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odessa, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Marcos, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita Falls, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morgantown, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Launceston, Tasmania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
- Belgium (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gilly
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haine-St.- Paul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Namur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turnhout
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barretos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newmarket, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- China (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sichuan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayonne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pierre-Bénite
- Germany (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hemer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Immenhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oldenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rheine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madurai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dublin, Ireland
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
- Portugal (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria da Feira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vila Franca de Xira
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elche
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., L'Hospitalet de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Majadahonda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terrassa
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fatih
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melikgazi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umuttepe
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edgbaston, Birmingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edinburgh, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester, United Kingdom

REFERENCES:
- [Derived] Govindan R, Senan S, Dickgreber N, Provencio M, Wu YL, Syrigos K, Parente B, Wilson M, Ziemiecki R, Chouaki N, Hossain A, San Antonio B, Winfree K, Vokes EE. Healthcare resource utilization and associated cost analysis of the PROCLAIM study in patients with stage III non-small-cell lung cancer. Curr Med Res Opin. 2019 Oct;35(10):1761-1767. doi: 10.1080/03007995.2019.1623185. Epub 2019 Jul 5. PMID 31125266
- [Derived] Brade AM, Wenz F, Koppe F, Lievens Y, San Antonio B, Iscoe NA, Hossain A, Chouaki N, Senan S. Radiation Therapy Quality Assurance (RTQA) of Concurrent Chemoradiation Therapy for Locally Advanced Non-Small Cell Lung Cancer in the PROCLAIM Phase 3 Trial. Int J Radiat Oncol Biol Phys. 2018 Jul 15;101(4):927-934. doi: 10.1016/j.ijrobp.2018.04.015. Epub 2018 Apr 12. PMID 29976505
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Started | 301 | 297
Received at Least One Dose of Study Drug | 283 | 272
Entered Consolidation Phase | 229 | 202
Completed | 177 (Study completion includes death due to any cause) | 180 (Study completion includes death due to any cause.)
Not Completed | 124 | 117
Not completed — Participants censored (no death events) | 124 | 117

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Arm A: Pemetrexed + Cisplatin and TRT: Participants were treated with Pemetrexed plus Cisplatin and concurrent TRT ("Concurrent Phase") for three 21-day cycles, followed by a 3-5 week "Recovery Period," then treated with consolidation chemotherapy with pemetrexed ("Consolidation Phase") for up to four 21-day cycles
  Concurrent Phase:
  Pemetrexed: 500 mg/m^2, IV on Day 1 of each 21-day cycle for 3 cycles. Cisplatin: 75 mg/m^2, IV on Day 1 of each 21-day cycle x 3 cycles. TRT: Beginning on Day 1 of chemotherapy, once daily fractions (2 Gy per day), 5 days a week for 6 weeks and 3 days to target 66 Gy in 33 fractions.
  Consolidation Phase:
  Pemetrexed: 500 mg/m^2, IV on Day 1 of each 21-day cycle up to 4 cycles
- Total: Total of all reporting groups
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT | Total
Number analyzed (Participants) | 301 | 297 | 598
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (9.6) | 58.5 (9.4) | 58.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 119 | 243
  Male | 177 | 178 | 355
Race/Ethnicity, Customized [Number; unit: participants]
  African | 15 | 12 | 27
  Caucasian | 217 | 204 | 421
  East Asian | 54 | 68 | 122
  Hispanic | 5 | 4 | 9
  Native American | 1 | 1 | 2
  West Asian | 6 | 6 | 12
  Missing (unknown) | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Argentina | 2 | 1 | 3
  United States | 58 | 76 | 134
  United Kingdom | 14 | 5 | 19
  Portugal | 7 | 11 | 18
  Spain | 38 | 27 | 65
  India | 14 | 14 | 28
  Greece | 13 | 3 | 16
  Canada | 16 | 10 | 26
  Netherlands | 26 | 20 | 46
  Turkey | 3 | 4 | 7
  Belgium | 21 | 23 | 44
  Ireland | 1 | 0 | 1
  China | 27 | 34 | 61
  Taiwan | 11 | 14 | 25
  Brazil | 7 | 9 | 16
  Korea, Republic of | 6 | 5 | 11
  Australia | 7 | 10 | 17
  France | 13 | 9 | 22
  Germany | 15 | 22 | 37
  Mexico | 2 | 0 | 2
ECOG performance status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status:
  0=Fully active, able to carry on all pre-disease performance without restriction
  1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, such as, light housework, office work
  participants
    0 | 148 | 145 | 293
    1 | 152 | 149 | 301
    Missing | 1 | 3 | 4
Disease stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIA - the cancer has spread to nearby tissue or spread to far away lymph nodes; Stage IIIB - cancer spread to opposite side of chest, more than one tumor within same lobe of lung.
  participants
    Stage IIIA | 140 | 142 | 282
    Stage IIIB | 161 | 152 | 313
    Missing | 0 | 3 | 3
Histology [Number; unit: participants]
  Adenocarcinoma | 226 | 226 | 452
  Large cell carcinoma | 16 | 21 | 37
  Other | 59 | 48 | 107
  Missing | 0 | 2 | 2
Smoking status [Number; unit: participants]
  Never smoked | 50 | 58 | 108
  Moderate smoker | 42 | 38 | 80
  Heavy smoker | 190 | 183 | 373
  Missing | 19 | 18 | 37
Baseline PET scan [Number; unit: participants] — Participant had a baseline Positron Emission Tomography (PET) scan for staging
  participants
    Yes | 250 | 241 | 491
    No | 51 | 56 | 107

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) time is from baseline to the date of death from any cause. For participants not known to have died as of the data cut-off date, OS time was censored at the last contact date the participant was known to be alive prior to the data cut-off date. OS was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to Date of Death from Any Cause (Up to 71.4 Months)
Population: All randomized participants. Arm A had 124 participants censored and Arm B had 117 participants censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Number analyzed (Participants) | 301 | 297
months | 26.81 [20.40 to 30.92] | 24.97 [22.18 to 29.83]
Statistical Analysis 1: Comparison: Arm A: Pemetrexed + Cisplatin and TRT vs Arm B: Etoposide + Cisplatin and TRT; Test type: Superiority or Other; p = 0.831, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.79 to 1.20]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) time is from baseline to the first date of documented objective progressive disease (PD) or death from any cause. For participants who were not known to have died or to have had objective PD as of the data inclusion cut-off date for a particular analysis, PFS was censored at the date of the last objective progression-free disease assessments. For participants who took any subsequent systemic anticancer therapy prior to progression or death, PFS was censored at the date of the last objective progression-free disease assessment prior to the start date of any subsequent systemic anticancer therapy. PFS time was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause (Up to 66.6 Months)
Population: All randomized participants. Arm A had 99 participants censored and Arm B had 87 participants censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Number analyzed (Participants) | 301 | 297
months | 11.37 [10.25 to 13.21] | 9.76 [8.38 to 11.73]
Statistical Analysis 1: Comparison: Arm A: Pemetrexed + Cisplatin and TRT vs Arm B: Etoposide + Cisplatin and TRT; Test type: Superiority or Other; p = 0.130, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.71 to 1.04]

3. Secondary Outcome: Objective Response Rate (Complete Response [CR] + Partial Response [PR])
Description: Overall response rate (ORR) is the best response of CR or PR as classified by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST, v1.1) guidelines. CR is defined as the disappearance of all target and non-target lesions, normalization of tumor marker level of non-target lesions, and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline to Measured Progressive Disease (Up to 7 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Number analyzed (Participants) | 301 | 297
percentage of participants | 35.9 [30.46 to 41.58] | 33.0 [27.67 to 38.66]
Statistical Analysis 1: Comparison: Arm A: Pemetrexed + Cisplatin and TRT vs Arm B: Etoposide + Cisplatin and TRT; Test type: Superiority or Other; p = 0.458, Log Rank

4. Other Pre Specified Outcome: Adverse Events: The Number of Deaths Per Treatment Group
Description: The number of deaths that occurred while on study drug, the number of deaths due to adverse events (AEs) while on study drug, and the number of deaths due to the study disease (that is, disease progression) while on study drug are presented. In addition, the number of deaths within 30 days of treatment discontinuation, the number of deaths due to AEs within 30 days of treatment discontinuation, and the number of deaths due to study disease within 30 days of treatment discontinuation are presented. For both the deaths due to AEs that occurred on study and for deaths due to AEs that occurred within 30 days of treatment discontinuation, the causality (events assess as possibly related [poss related] to study drug per investigator judgement) is also presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 30 Days Post Study
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Number analyzed (Participants) | 283 | 272
participants
  On study drug (total) | 12 | 6
  On study drug: Due to AE | 10 | 4
  On study drug: Due to AE poss related | 5 | 3
  On study drug: Due to study disease | 2 | 0
  Within 30 Days of Discontinuation (disc) (total) | 10 | 6
  Within 30 Days of Disc: Due to AE | 5 | 4
  Within 30 Days of Disc: Due to AE poss related | 2 | 0
  Within 30 Days of Disc: Due to study disease | 5 | 2

5. Secondary Outcome: Survival Rates at 1, 2, and 3 Years
Description: The probability that survival time is at least 1, 2, or 3 years was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to Date of Death from Any Cause (Up to 71.4 Months)
Population: All randomized participants. Arm A had 124 participants censored and Arm B had 117 participants censored.
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Number analyzed (Participants) | 301 | 297
probability of survival
  1 year (12 months) | 0.76 [0.70 to 0.80] | 0.77 [0.72 to 0.81]
  2 years (24 months) | 0.52 [0.46 to 0.58] | 0.52 [0.46 to 0.58]
  3 years (36 months) | 0.40 [0.34 to 0.46] | 0.37 [0.31 to 0.43]

6. Secondary Outcome: First Site of Disease Failure in Terms of Relapse
Description: The percentage of participants with first sites of disease failure in terms of relapse within the radiation treatment field, inside the thorax, (outside of the radiation field), or distant disease are presented. Results were summarized using Kaplan-Meier estimates. Some participants relapsed in more than 1 location/site and appear in more than a single category.
Time Frame: Baseline to Relapse (Up to 66.6 Months)
Population: All randomized participants with objective PD.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Number analyzed (Participants) | 166 | 190
percentage of participants
  Relapsed within the radiation treatment field | 37.3 [30.0 to 45.2] | 45.8 [38.6 to 53.2]
  Relapsed inside thorax, outside of radiation field | 20.5 [14.6 to 27.4] | 16.3 [11.4 to 22.4]
  Relapsed distant disease | 50.0 [42.2 to 57.8] | 45.8 [38.6 to 53.2]
Statistical Analysis 1: Comparison: Arm A: Pemetrexed + Cisplatin and TRT vs Arm B: Etoposide + Cisplatin and TRT; Relapsed within the radiation treatment field; Test type: Superiority or Other; p = 0.132, Fisher Exact
Statistical Analysis 2: Comparison: Arm A: Pemetrexed + Cisplatin and TRT vs Arm B: Etoposide + Cisplatin and TRT; Relapsed inside thorax, outside of radiation field; Test type: Superiority or Other; p = 0.337, Fisher Exact
Statistical Analysis 3: Comparison: Arm A: Pemetrexed + Cisplatin and TRT vs Arm B: Etoposide + Cisplatin and TRT; Relapsed distant disease; Test type: Superiority or Other; p = 0.457, Fisher Exact

7. Secondary Outcome: Percentage of Participants With a Post Baseline Swallowing Diary Score >=4
Description: Participants were provided with a swallowing diary to record issues with swallowing using a 5-point categorical scale: (1) no problems; (2) mild soreness; (3) swallowing solids with some difficulty; (4) inability to swallow solids; and (5) inability to swallow liquids. Participants rated swallowing over the previous 24 hours. The percentage of participants was calculated by dividing the number of with a post baseline swallowing diary score >=4 by total number of participants analyzed, multiplied by 100. No adjustments were made for the number of available assessments nor were any interpolation of missing assessments made.
Time Frame: Baseline through 30 Days Post Study
Population: All randomized participants with at least one post baseline swallowing diary score.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pemetrexed + Cisplatin and TRT | Arm B: Etoposide + Cisplatin and TRT
Number analyzed (Participants) | 284 | 269
percentage of participants | 33.8 [26.7 to 37.5] | 29.0 [21.3 to 31.7]
Statistical Analysis 1: Comparison: Arm A: Pemetrexed + Cisplatin and TRT vs Arm B: Etoposide + Cisplatin and TRT; Test type: Superiority or Other; p = 0.150, Fisher Exact

ADVERSE EVENTS:
Description: Randomized participants who received at least one dose of study drug.
Groups:
- Arm A:: Arm A: Participants were treated with pemetrexed plus cisplatin and concurrent thoracic radiation TRT ("Concurrent Phase") for three 21-day cycles, followed by a 3-5 week "Recovery Period," then treated with consolidation chemotherapy with pemetrexed ("Consolidation Phase") for four 21-day cycles
  Concurrent Phase:
  Pemetrexed: 500 mg/m^2, IV on Day 1 of each 21-day cycle for 3 cycles. Cisplatin: 75 mg/m^2, IV on Day 1 of each 21-day cycle x 3 cycles. TRT: Beginning on day 1 of chemotherapy, once daily fractions (2 Gy per day), 5 days a week for 6 weeks and 3 days to target 66 Gy in 33 fractions.
  Consolidation Phase:
  Pemetrexed 500 mg/m^2, IV on Day 1 of each 21-day cycle up to 4 cycles.
- Arm B: Etoposide + Cisplatin and TRT: Participants were treated with Etoposide plus Cisplatin and concurrent TRT ("Concurrent Phase") for two 28-day cycles, followed by a 3-5 week "Recovery Period," then received consolidation treatment with cytotoxic chemotherapy of choice ("Consolidation Phase") for up to 2 cycles
  Concurrent Phase:
  Etoposide/Cisplatin (28-day cycle); Etoposide: 50 mg/m^2, IV on Days 1 to 5 and Days 29 to 33 and Cisplatin: 50 mg/m^2, IV on Days1, 8, 29, and 36
  Consolidation Phase options:
  Option 1: Continue the same treatment plan as Concurrent Phase
Arm/Group | Arm A: | Arm B: Etoposide + Cisplatin and TRT
Serious Adverse Events (participants affected / at risk) | 134/283 | 145/272
Other Adverse Events (participants affected / at risk) | 279/283 | 269/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (N=283) | Arm B: Etoposide + Cisplatin and TRT (N=272)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 5 (22)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (14) | 24 (25)
Leukopenia (Blood and lymphatic system disorders) | 4 (6) | 6 (12)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (11)
Neutropenia (Blood and lymphatic system disorders) | 8 (21) | 13 (16)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4) | 5 (7)
Atrial fibrillation (Cardiac disorders) | 4 (11) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Endocarditis noninfective (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 2 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 1 (9)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Aplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (11)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aorto-oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (15) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (8) | 5 (7)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (7) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (27) | 7 (14)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (16)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 26 (63) | 29 (89)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 14 (23) | 8 (9)
Asthenia (General disorders) | 2 (4) | 1 (1)
Chest pain (General disorders) | 3 (5) | 5 (5)
Death (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (4) | 4 (9)
Malaise (General disorders) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 1 (4) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (10)
Pain (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 11 (14) | 4 (6)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2)
Device related infection (Infections and infestations) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Infectious colitis (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (7) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (4) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 18 (30) | 18 (32)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (3)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (2) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (6) | 2 (2)
Sepsis (Infections and infestations) | 1 (2) | 4 (5)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (6) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation fibrosis - lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 7 (18) | 13 (20)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 7 (19) | 5 (13)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (3) | 1 (14)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (4) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 3 (5)
Weight decreased (Investigations) | 4 (13) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (8) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 7 (15) | 6 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (17)
Lung infiltration malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (17) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (2) | 1 (11)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (4) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (7) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (3) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (19) | 3 (19)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 10 (14)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (15)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (4) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 2 (6)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (2)
Thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (N=283) | Arm B: Etoposide + Cisplatin and TRT (N=272)
Anaemia (Blood and lymphatic system disorders) | 88 (336) | 94 (312)
Leukopenia (Blood and lymphatic system disorders) | 63 (267) | 71 (237)
Lymphopenia (Blood and lymphatic system disorders) | 62 (297) | 47 (170)
Neutropenia (Blood and lymphatic system disorders) | 92 (252) | 123 (359)
Thrombocytopenia (Blood and lymphatic system disorders) | 39 (116) | 53 (132)
Tinnitus (Ear and labyrinth disorders) | 15 (40) | 8 (27)
Abdominal pain upper (Gastrointestinal disorders) | 35 (94) | 8 (13)
Constipation (Gastrointestinal disorders) | 112 (312) | 129 (284)
Diarrhoea (Gastrointestinal disorders) | 55 (88) | 63 (104)
Dyspepsia (Gastrointestinal disorders) | 43 (148) | 37 (95)
Dysphagia (Gastrointestinal disorders) | 140 (567) | 110 (317)
Nausea (Gastrointestinal disorders) | 175 (532) | 144 (365)
Odynophagia (Gastrointestinal disorders) | 24 (103) | 23 (56)
Oesophagitis (Gastrointestinal disorders) | 119 (470) | 99 (253)
Stomatitis (Gastrointestinal disorders) | 26 (50) | 12 (23)
Vomiting (Gastrointestinal disorders) | 110 (244) | 95 (173)
Asthenia (General disorders) | 64 (249) | 35 (101)
Chest pain (General disorders) | 40 (154) | 32 (71)
Fatigue (General disorders) | 139 (685) | 131 (472)
Mucosal inflammation (General disorders) | 31 (73) | 23 (64)
Oedema peripheral (General disorders) | 24 (61) | 12 (28)
Pyrexia (General disorders) | 56 (76) | 42 (60)
Pneumonia (Infections and infestations) | 17 (36) | 12 (21)
Upper respiratory tract infection (Infections and infestations) | 15 (29) | 11 (18)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 16 (50) | 18 (42)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 22 (52) | 16 (29)
Radiation skin injury (Injury, poisoning and procedural complications) | 45 (159) | 37 (81)
Alanine aminotransferase increased (Investigations) | 21 (84) | 11 (25)
Aspartate aminotransferase increased (Investigations) | 20 (63) | 9 (18)
Blood creatinine increased (Investigations) | 26 (67) | 16 (32)
Haemoglobin decreased (Investigations) | 48 (218) | 43 (155)
Neutrophil count decreased (Investigations) | 32 (115) | 31 (76)
Platelet count decreased (Investigations) | 24 (74) | 33 (78)
Weight decreased (Investigations) | 69 (257) | 61 (204)
White blood cell count decreased (Investigations) | 47 (212) | 43 (131)
Decreased appetite (Metabolism and nutrition disorders) | 104 (366) | 88 (228)
Dehydration (Metabolism and nutrition disorders) | 19 (31) | 24 (38)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (57) | 8 (25)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (43) | 32 (49)
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 (84) | 32 (84)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (52) | 22 (55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (33) | 17 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (94) | 21 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (41) | 11 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (26) | 14 (30)
Dizziness (Nervous system disorders) | 50 (152) | 45 (96)
Dysgeusia (Nervous system disorders) | 31 (122) | 22 (60)
Headache (Nervous system disorders) | 36 (92) | 34 (67)
Neuropathy peripheral (Nervous system disorders) | 14 (35) | 25 (64)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (80) | 21 (61)
Anxiety (Psychiatric disorders) | 17 (61) | 12 (35)
Insomnia (Psychiatric disorders) | 52 (175) | 42 (126)
Cough (Respiratory, thoracic and mediastinal disorders) | 105 (430) | 84 (273)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 93 (308) | 53 (142)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 31 (84) | 17 (33)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 (43) | 24 (41)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 23 (59) | 8 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (110) | 103 (389)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (52) | 15 (43)
Erythema (Skin and subcutaneous tissue disorders) | 17 (50) | 13 (29)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (55) | 11 (19)
Rash (Skin and subcutaneous tissue disorders) | 45 (110) | 40 (93)
Hypotension (Vascular disorders) | 3 (6) | 16 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days